CLINICAL TRIAL: NCT00830570
Title: in Typical Community Practice Settings
Brief Title: The Clinical and Economic Impact of Pharmacogenomic Testing of Warfarin Therapy in Typical Community Practice Settings
Acronym: MHSMayoWarf1
Status: Completed | Type: Observational
Sponsor: Medco Health Solutions, Inc. (Industry)
Collaborators: Mayo Clinic (Other); Washington University School of Medicine (Other)
Responsible Party: Robert Epstein, MD, MS, Medco Health Solutions, Inc.
Other Study IDs: MedcoWarfarin1
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Embolism and Thrombosis; Embolism; Vascular Diseases; Warfarin; Venous Thromboembolism; Thrombosis; Thromboembolism
Keywords: CYP2C9; VKORC1; polymorphism; warfarin; Coumadin
MeSH Terms: conditions — Embolism and Thrombosis; Embolism; Vascular Diseases; Venous Thromboembolism; Thrombosis; Thromboembolism; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2 | interventions — Warfarin; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw and buccal swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Historical control group. Patients in this group are drawn from the same plan populations as the intervention group, but they are identified during the 1-year period prior to the start of patient enrollment in the intervention group. The historical control group is closely matched with the intervention group on demographic characteristics, practice patterns, and benefit plan features that may affect resource utilization.
- 2: Concurrent control group. Patients in this group are drawn from different set of plan populations, but they initiate warfarin treatment during the same time period as patients in the intervention group. Outcomes data for the concurrent control group will be used to evaluate whether any differences between the intervention group and the historical control group can be attributed to changes in clinical practice over time. Baseline data for the concurrent control group will help validate the incidence assumptions used in the calculation of statistical power. This use of baseline population norms is an effective means of limiting bias in quasi-experimental studies.
- 3: Active study group. For plans participating in the active arm of the study, enrollment is offered to every patient who initiates warfarin therapy during the enrollment period (beginning in July 2007) and who meets the eligibility criteria. Patients are identified for the active study group if they have a warfarin pharmacy claim and no prior warfarin claims during the preceding 180 days. Only patients who remain eligible for the pharmacy benefit throughout the study period are included in the final sample.
  Interventions: Other: CYP 2C9 and VKORC1 Testing for Warfarin

INTERVENTIONS:
Other: CYP 2C9 and VKORC1 Testing for Warfarin — Test patients for their warfarin sensitivity and provide this information to their physician authorizing the test.
  Other Names: Genetic testing for drug sensitivity
  Groups: 3

SUMMARY:
The purpose of this quasi-experiment study, which could also be classified as a prospective observational intervention study, is to assess the impact of cytochrome P450 2C9 (CYP 2C9) and vitamin K epoxide reductase complex, subunit 1 (VKORC1) testing within a primary patient care setting.

DETAILED DESCRIPTION:
Anticoagulation therapy with warfarin is the most common mode of treatment and prophylaxis for venous and arterial thromboembolic conditions. Warfarin is metabolized in the liver by the cytochrome P450 system, the cytochrome P450 2C9 (CYP 2C9) isoenzyme specifically, and polymorphisms in the CYP 2C9 gene have been associated with changes in metabolic function of the translated isoenzyme . These polymorphisms result in reduced metabolism of warfarin as compared to subjects having the wild type gene, consequently leading to systemic accumulation of warfarin; it is theorized that this leads to higher risk of adverse events. Other allelic variations have also been linked to changes in vitamin K conservation through their effects on vitamin K epoxide reductase complex, subunit 1 (VKORC1) . The combined impact of CYP 2C9 and VKORC1 polymorphisms on warfarin's pharmacology have recently been reported.

It is hypothesized that evaluation of genomic allelic type guided warfarin dosing will reduce thromboembolic and bleeding risks associated with warfarin therapy, and that adoption of a genetic testing strategy in a primary patient care setting would improve warfarin effectiveness and patient safety, and reduce costs to health care payers.

ELIGIBILITY:
Inclusion Criteria:

* Female and male age range of 40-75
* Patients who are in the induction phase of warfarin
* Patients receiving warfarin to prevent or treat thromboembolic conditions (e.g., post orthopedic surgery prophylaxis, deep venous thrombosis, atrial fibrillation, pulmonary embolism, heart failure)
* Patient willing to provide informed consent prior to the specimen collection procedure
* Patient whose physician is willing to order the genetic test

Exclusion Criteria:

* Age < 40 or > 75
* Previous use of warfarin within 180 days of initiating new warfarin therapy
* Hospitalized for seven or more days before first claim for warfarin
* Previous history of genetic testing for warfarin therapy
* Known hypersensitivity to warfarin
* Patient or physician refusal to participate in the study
* Patients using warfarin residing in Olmsted County, MN

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The active study population consists of male and female covered lives with Medco for clients have agreed to enroll their members for ages 40-75 for new warfarin starts who match the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1635 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to determine whether the addition of genotyping to usual care will reduce the hospitalization rates for hemorrhage or thromboembolism related to warfarin use during the first 6 months of treatment. | 6 months

SECONDARY OUTCOMES:
The secondary objective is to determine physician and patient acceptance of the technology. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Epstein, MD, MS, Principal Investigator — Medco Health Solutions, Inc.
Locations (1):
- Medco Health Solutions, Inc., Franklin Lakes, New Jersey, United States

REFERENCES:
- [Result] Epstein RS, Moyer TP, Aubert RE, O Kane DJ, Xia F, Verbrugge RR, Gage BF, Teagarden JR. Warfarin genotyping reduces hospitalization rates results from the MM-WES (Medco-Mayo Warfarin Effectiveness study). J Am Coll Cardiol. 2010 Jun 22;55(25):2804-12. doi: 10.1016/j.jacc.2010.03.009. Epub 2010 Apr 8. PMID 20381283